CLINICAL TRIAL: NCT05127512
Title: Pelvic Floor Disorder Education in the Prenatal Period, a Randomized Controlled Trial
Brief Title: Pelvic Floor Disorder Education in Prenatal Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Chandhana Paka, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY-20-03435
Record Dates: First submitted 2021-10-28; First posted 2021-11-19 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Pelvic Floor Disorders
Keywords: Pelvic floor disorders; Education; Prenatal education; Video education
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Control participants will only complete the knowledge questionnaire in addition to a non-validated survey created by the investigators to collect demographic information as well as attitudes towards treatments of pelvic floor disorders.
- Video Group (Experimental): These participants will be administered the study intervention, which entails viewing an education video on pelvic floor disorders.
  Interventions: Other: Education Video

INTERVENTIONS:
Other: Education Video — A 6.47-minute education video was created by the research group based on American Urogynecology Society (AUGS) and International Urogynecologic Association (IUGA) patient education pamphlets. Participants in the intervention group will be asked to watch this video after completing a baseline knowledge questionnaire of pelvic floor disorders.
  Arms: Video Group

SUMMARY:
Pelvic floor disorders (PFDs) are common conditions that can have significant impacts on patients' quality of life and psychosocial well-being. It is well known that patients who have experienced pregnancy and childbirth are at risk of developing these conditions, either during pregnancy, postpartum, or later in life. However, many women are unaware of this predisposing risk factor. Additionally, overall knowledge of these conditions is low in both the general and obstetrics population.

Video education has been used in various fields with success in improving patient knowledge of specific topics and conditions. To the researchers' knowledge, no studies have evaluated this modality for educating obstetrics patients on PFDs. The aim of this study is to determine whether the use of an educational video will improve knowledge of PFDs compared to routine prenatal counseling, using a validated knowledge questionnaire.

DETAILED DESCRIPTION:
Once verbal consent is obtained, participants will be randomly assigned in a 1:1 ratio to the intervention (video education) or control group (routine prenatal visit only). Group assignments will be performed using computer-generated randomization. All participants will complete a paper questionnaire including basic demographic information, prior history of pelvic floor disorders, and current PFD symptoms. Participants assigned to the routine prenatal visit only will be instructed to complete the Prolapse and Incontinence Knowledge Questionnaire (PIKQ). The PIKQ is a validated 24-item questionnaire designed to assess knowledge of PFDs, including two 12-item subscales on urinary incontinence (PIKQ-UI) and prolapse (PIKQ-POP).

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older in their third trimester of pregnancy (37 weeks of gestation or greater)
* English-speaking

Exclusion Criteria:

* Non-English-speaking patients
* Gestational age < 37 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 94 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Change in Prolapse and Incontinence Knowledge Questionnaire | Baseline, 1 day ( the time of enrollment) and at 6-8 weeks
  The questionnaire is divided into two separate 12-item subscales on urinary incontinence (PIKQ-UI) and prolapse (PIKQ-POP). Subscales from 0 to 12. Total scale from 0-24. A higher score indicates higher proficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Chandhu Paka, MD, Principal Investigator — Mount Sinai West
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. For individual participant data meta-analysis. Proposals should be directed to bhgaigbe@gmail.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website tbd.

REFERENCES:
- [Background] Wu JM, Matthews CA, Conover MM, Pate V, Jonsson Funk M. Lifetime risk of stress urinary incontinence or pelvic organ prolapse surgery. Obstet Gynecol. 2014 Jun;123(6):1201-1206. doi: 10.1097/AOG.0000000000000286. PMID 24807341
- [Background] Hyakutake MT, Han V, Cundiff GW, Baerg L, Koenig NA, Lee T, Geoffrion R. Pelvic Floor Health Education: Can a Workshop Enhance Patient Counseling During Pregnancy? Female Pelvic Med Reconstr Surg. 2016 Sep-Oct;22(5):336-9. doi: 10.1097/SPV.0000000000000285. PMID 27171319
- [Background] Geoffrion R, Robert M, Ross S, van Heerden D, Neustaedter G, Tang S, Milne J. Evaluating patient learning after an educational program for women with incontinence and pelvic organ prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Oct;20(10):1243-52. doi: 10.1007/s00192-009-0919-5. Epub 2009 Jun 11. PMID 19517050
- [Background] Howell EA. Lack of patient preparation for the postpartum period and patients' satisfaction with their obstetric clinicians. Obstet Gynecol. 2010 Feb;115(2 Pt 1):284-289. doi: 10.1097/AOG.0b013e3181c8b39b. PMID 20093900
- [Background] Liu J, Tan SQ, Han HC. Knowledge of pelvic floor disorder in pregnancy. Int Urogynecol J. 2019 Jun;30(6):991-1001. doi: 10.1007/s00192-019-03891-3. Epub 2019 Feb 19. PMID 30783706